CLINICAL TRIAL: NCT03728985
Title: Evaluation of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis in the Treatment of Thoracoabdominal and Pararenal Aortic Aneurysms
Acronym: TAMBE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAA 17-01
Expanded Access: NCT05442489 (Approved for marketing)
Record Dates: First submitted 2018-09-28; First posted 2018-11-02 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Thoracoabdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Intervention Model Description: This study contains two single arm substudies. A primary study arm and a secondary study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Primary Study Arm (Active Comparator): TAAA requiring only TAMBE System. Crawford Type IV TAAA and Pararenal (n= 102)
  Interventions: Device: GORE EXCLUDER Thoracoabdominal Branch Endoprosthesis
- Secondary Study Arm (Experimental): TAAA requiring TAMBE System and CTAG Device(s). Crawford Type I-III (n= 20 - 100)
  Interventions: Device: GORE EXCLUDER Thoracoabdominal Branch Endoprosthesis

INTERVENTIONS:
Device: GORE EXCLUDER Thoracoabdominal Branch Endoprosthesis — Endovascular Aortic Stent-Graft
  Other Names: TAMBE

SUMMARY:
Prospective, non-randomized, , multicenter study with two independent arms:

* Primary Study Arm - TAAA and Pararenal aneurysms requiring only TAMBE System. Hypothesis-driven analysis.

  * Up to 65 additional subjects may be implanted in Continued Access Phase under the Primary Study Arm only
* Secondary Study Arm - TAAA requiring TAMBE System and CTAG Device(s). Non hypothesis-driven analysis.

Minimum: 122 implanted subjects. Maximum: 202 implanted subjects with up to 65 additional subjects implanted in Continued Access (Primary Study arm)

ELIGIBILITY:
Inclusion Criteria:

1. Aortic aneurysm involving the visceral vessels requiring treatment defined as at least one of the following:

   * Fusiform aneurysm diameter ≥ 5 cm
   * Saccular aneurysm (no diameter requirement)
   * Rapid aneurysm growth (≥ 5 mm in one year)
2. Aortic aneurysm that involves the abdominal aorta, with:

   * Involvement of at least one visceral vessel and aneurysmal extension as far as 65 mm proximal to the celiac artery, and/or
   * No normal aorta between the upper extent of aneurysm and renal artery(s)
3. Adequate access for TAMBE Device components (femoral, axillary, and / or brachial arteries as required)
4. Age ≥ 19 years at the time of informed consent signature
5. Male or infertile female
6. Patient assessment favors an endovascular approach when compared to open surgical repair, as deemed by the treating physician
7. Capable of complying with protocol requirements, including follow-up
8. An Informed Consent Form signed by Subject or legal representative
9. Sufficient distal landing zones in both iliac arteries, with at least one patent internal iliac artery and without planned placement of a branched iliac device, or planned coverage/occlusion/embolization of any patent internal iliac artery.
10. Appropriate aortic anatomy to receive the TAMBE Device defined as all of the following:

    * For the TAMBE aortic component, proximal aortic landing zone diameters between 22-34 mm
    * Proximal seal zone ≥ 20 mm in length
    * Aortic neck angle ≤ 60°
    * Distal landing zone (iliac arteries) 8-25 mm
    * Distal seal zone in iliac arteries of at least 10 mm in length
    * Renal artery landing zone diameters between 4-10 mm
    * Celiac and superior mesenteric artery landing zone diameters between 5-12 mm
    * ≥ 15 mm landing zone in each branch vessel
    * Landing zones in the proximal and distal aorta and all branch vessels cannot be aneurysmal, heavily calcified, or heavily thrombosed
    * Patent left subclavian artery

    Secondary Study Arm Only:
11. If aneurysm extends greater than 65 mm above celiac artery, proximal extension with a CTAG Device is required. The aortic landing zone diameter treatment range with the CTAG Device is 19.5-32 mm
12. The most proximal aspect of the aneurysm is at least 2.0 cm distal to the left subclavian artery.
13. The most proximal aortic device seal zone will be within native aorta or a previously-deployed TAG or CTAG Device • Placement inside a Dacron graft or another device manufacturer's stent graft will not be supported

Exclusion Criteria:

The patient is / has:

1. Prior open, aortic surgery of the ascending aorta or aortic arch
2. Ruptured or leaking aortic aneurysm
3. Aneurysmal dilatation due to chronic aortic dissection
4. Infected aorta
5. Mycotic aneurysm
6. Life expectancy <2 years
7. Myocardial infarction or stroke within 1 year of treatment (staged or index procedure)
8. Systemic infection which may increase risk of endovascular graft infection
9. Degenerative connective tissue disease, e.g. Marfan's or Ehler-Danlos Syndrome
10. Participation in an investigational drug study (within 30 days of last administration) or investigational medical device study (within 1 year of implant) from the time of study screening
11. History of drug abuse, e.g. cocaine or amphetamine or alcohol, within 1 year of treatment
12. Tortuous or stenotic iliac and / or femoral arteries and the inability to use a conduit for vascular access
13. A branch vessel(s) that is dissected or has significant calcification, tortuosity, thrombus formation that would interfere with device delivery or ability to exclude from blood flow
14. Known sensitivities or allergies to the device materials
15. Previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or known hypersensitivity to heparin
16. Patient has body habitus or other medical condition which prevents adequate fluoroscopic and CT visualization of the aorta
17. Renal Insufficiency (creatinine value > 1.8 mg/dL, GFR < 30, or patient undergoing dialysis)
18. Known concomitant aneurysm of the ascending aorta or aortic arch anticipated to require surgical intervention within one year of study treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2026-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Farber, MD, Principal Investigator — University of North Carolina
Locations (44):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Keck Medical Center of USC, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente San Francisco Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - MedStar Health Research Institute - MedStar Washington Hospital, Washington D.C., District of Columbia
  - University of Florida - Gainesville, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan - Cardiac Surgery, Ann Arbor, Michigan
  - Essentia Health, Duluth, Minnesota
  - Division of Vascular Surgery - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Mount Sinai West, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Sanger Heart & Vascular Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPP Heart and Vascular Institute, Pittsburgh, Pennsylvania
  - University of Tennessee -University Vascular Surgeons, Knoxville, Tennessee
  - St. David's Healthcare, Austin, Texas
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The Methodist Hospital - Houston, Houston, Texas
  - University of Texas Health Science Center, Houston, Texas
  - Sentara Medical Group, Norfolk, Virginia
  - Carilion Clinic Hospitals, Roanoke, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Aurora Health Care, Metro Inc., Milwaukee, Wisconsin
- United Kingdom (2):
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - St. Mary's Hospital, Imperial College Healthcare, NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects went through Screening after Enrollment. Subjects available and eligible for Primary Arm were implanted.
Period: Overall Study
Arm/Group | Primary Study Arm
Started | 102
Primary Endpoint Determined | 102 (Subjects with at least one Primary Endpoint determined)
Completed | 102 (Subjects with 12 month follow-up or both co-primary endpoints determined)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (3.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity only collected for subjects in the US
  Participants
    number analyzed (Participants) | 99
    Hispanic or Latino | 2
    Not Hispanic or Latino | 92
    Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Subject Race is only collected for the subjects in the US
  Participants
    number analyzed (Participants) | 99
    American Indian or Alaska Native | 2
    Asian | 4
    Native Hawaiian or Other Pacific Islander | 1
    Black or African American | 4
    White | 84
    More than one race | 0
    Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 99
  United Kingdom | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With Uncomplicated Technical Success and Freedom From Procedural Safety Composite Event
Description: Percent of Subjects with Device Technical Success Composite Event and freedom from Procedural Safety Composite Event.
  Device Technical Success Composite Events during Index Procedure:
  Successful Access and Delivery Successful and Accurate Deployment Successful Withdrawal
  Procedural Safety during 30 days of Index Procedure:
  Stented Segment Aortic Rupture Lesion-Related Mortality Permanent Paraplegia Permanent Paraparesis New Onset Renal Failure Requiring Dialysis Severe Bowel Ischemia Disabling Stroke
Time Frame: From start of Index Procedure to 59 Days Post Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
Participants
  Subjects with Device Tech Success and Freedom from Procedural Safety Event (Index Proc to 59 Days) | 79
  Failure of Device Uncomplicated Technical Success (During Index Procedure) | 19
  Failure of Successful Access and Delivery(During Index Procedure) | 0
  Failure of Successful and Accurate Deployment(During Index Procedure) | 19
  Deployment/Kink/Twist/Obst/planned location(During Index Procedure) | 1
  Unplanned Placement of Non-TAMBE(During Index Procedure) | 19
  Use of Non-TAMBE to correct Iatrogenic(During Index Procedure) | 4
  Failure of Successful Withdrawal(During Index Procedure) | 0
  Procedural Safety Events (Index Procedure to 59 Days) | 8
  Stented Segment Aortic Rupture (Index Procedure to 59 Days) | 1
  Lesion Related Mortality(Index Procedure to 59 Days) | 0
  Permanent Paraplegia(Index Procedure to 59 Days) | 2
  Permanent Paraparesis(Index Procedure to 59 Days) | 3
  New Onset Renal Failure Requiring Dialysis(Index Procedure to 59 Days) | 2
  Severe Bowel Ischemia(Index Procedure to 59 Days) | 0
  Disabling Stroke(Index Procedure to 59 Days) | 1
Statistical Analysis 1: Comparison: Primary Study Arm; Test type: Non-Inferiority — Performance Goal 80%; p = 0.5908, Fisher Exact; Absolute Percentage with Success = 77.5, 90% CI 2-sided [69.6 to 84.1] — The lower estimated confidence interval above the Performance Goal of 80% would be considered success

2. Primary Outcome: Percent of Subjects Free From Clinically Significant Reintervention / Lesion-Related Mortality
Description: Composite Outcome of Lesions-Related Mortality and Clinically Significant Reinterventions through 12 Months for Pre-defined Reasons.
Time Frame: 12 Months
Population: Subjects not available for assessment at 12 months were excluded from the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
Participants
  Freedom from Clinically Sig. Reintervention and Lesion Related Mortality Through 12 Months: number analyzed (Participants) | 84
  Freedom from Clinically Sig. Reintervention and Lesion Related Mortality Through 12 Months | 60
  Clinically Significant Reintervention Through 12 Months: number analyzed (Participants) | 85
  Clinically Significant Reintervention Through 12 Months | 25
  Clinically-Indicated Condition: number analyzed (Participants) | 81
  Clinically-Indicated Condition | 6
  Untreated Device Seal Zone Endoleak: number analyzed (Participants) | 82
  Untreated Device Seal Zone Endoleak | 0
  Target-Lesion Growth > 5mm: number analyzed (Participants) | 84
  Target-Lesion Growth > 5mm | 5
  Rupture: number analyzed (Participants) | 94
  Rupture | 1
  Failure of Device Effectiveness (Compromise Device Seal Zone/Integrity2): number analyzed (Participants) | 94
  Failure of Device Effectiveness (Compromise Device Seal Zone/Integrity2) | 7
  Patient Safety Events (Total Occlusion of Device component2): number analyzed (Participants) | 95
  Patient Safety Events (Total Occlusion of Device component2) | 14
  Complicated Device System Prophylaxis (RI req Hospitalization2): number analyzed (Participants) | 95
  Complicated Device System Prophylaxis (RI req Hospitalization2) | 4
  Lesion Related Mortality Through 12 Months: number analyzed (Participants) | 94
  Lesion Related Mortality Through 12 Months | 0
Statistical Analysis 1: Comparison: Primary Study Arm; Test type: Non-Inferiority — Performance Goal 68%; p = 0.7017, Fisher Exact; Percentage with Success = 70.6, 90% CI 2-sided [61.4 to 78.7]

3. Secondary Outcome: Percent of Subjects With Aneurysm-related Mortality
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
Participants | 0

4. Secondary Outcome: Percent of Subjects With Stented Segment Aortic Rupture
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
Participants | 1

5. Secondary Outcome: Percent of Subjects With Lesion Related Mortality
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
Participants | 0

6. Secondary Outcome: Percent of Subjects With Permanent Paraplegia
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
Participants | 2

7. Secondary Outcome: Percent of Subjects With Permanent Paraparesis
Time Frame: 30 days of index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
Participants | 3

8. Secondary Outcome: Percent of Subjects With New Onset Renal Failure Requiring Dialysis
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
Participants | 2

9. Secondary Outcome: Percent of Subjects With Severe Bowel Ischemia
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
Participants | 0

10. Secondary Outcome: Percent of Subjects With Disabling Stroke
Description: Stroke will be assessed using the Modified Rankin Scale. Stroke identified as having occurred within 30 days of the index endovascular procedure, combined with mRS ≥2 with an increase from baseline of at least one grade at 90 days.
  Modified Rankin Scale:
  0 - No Symptoms
  1. No significant disability. Able to carry out all usual activities, despite some symptoms
  2. Slight Disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. Moderate Disability. Requires some help, but able to walk unassisted
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe Disability. Requires constant nursing care and attention, bedridden, incontinent
  6. Dead
  Higher Values are worse. A total score will not be computed, but a change from baseline will be calculated as (90 Day Post-Stroke MRS Score - Baseline MRS Score)
Time Frame: 120 days (30 Days for Initial Stroke, plus 90 Days for Followup MRS Score)
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
Participants | 1

11. Secondary Outcome: Percent of Subjects With Access-Related Complications
Time Frame: 30 days of index procedure
Reporting Status: Not Posted

12. Secondary Outcome: Mean Procedural Blood Loss at Index Procedure
Time Frame: Index Procedure
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
ml | 299.9 (295.5)

13. Secondary Outcome: Procedure Time
Time Frame: Index Procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
minutes | 315.3 (103.3)

14. Secondary Outcome: Length of Hospital Stay
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 102
days | 4.9 (3.45)

15. Secondary Outcome: Percent of Subjects With Extended Technical Clinical Success
Description: Patients who present within the 30-Day follow-up with no Type I or Type III endoleak, as evaluated by CTA, and free from device-related intervention.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 93
Participants | 0

16. Secondary Outcome: Percent of Subjects With Type I Endoleak
Description: Endoleak arising from the proximal or distal sealing zone of a device perfusing the aneurysm
  * Type IA: Inadequate seal at the proximal end of the device placed in the aorta
  * Type IB: Inadequate seal at the distal end of the device placed in iliac vessel
  * Type IC: Inadequate seal at the distal end of a device placed inside branch vessel Reported as ratio with the number of subjects with Type I Endoleak as numerator, number of subjects with an evaluable result as denominator. Ratios of Type IA, IB, and IC will also be reported.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 81
Participants | 0

17. Secondary Outcome: Percent of Subjects With Type II Endoleak
Description: Endoleak arising from a patent branch vessel perfusing the aneurysm, e.g., lumbar or inferior mesenteric branch.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 91
Participants | 64

18. Secondary Outcome: Percent of Subjects With Type III Endoleak
Description: Type III Endoleak through 12 months - Endoleak arising from the component junction(s) of the prosthesis or due to damage to the graft material perfusing the aneurysm.
  * Type III General: A Type III endoleak whose source cannot be differentiated between an intercomponent junction or graft tear
  * Type IIIA: Modular disconnection or apposition failure
  * Type IIIB: Graft tear
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 81
Participants | 0

19. Secondary Outcome: Percent of Subjects With Type IV Endoleak
Description: Endoleak of whole blood through the graft fabric perfusing the aneurysm
  Reported as a ratio. Numerator: Number of Subjects with Type IV Endoleak. Denominator: Number of Subjects with an Evaluable Result
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 81
Participants | 0

20. Secondary Outcome: Percent of Subjects With Type IV Indeterminate Endoleak
Description: Endoleak perfusing the aneurysm without a definitive source
  Reported as a ratio. Numerator: Number of Subjects with Type IV Endoleak. Denominator: Number of Subjects with an Evaluable Result
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 84
Participants | 14

21. Secondary Outcome: Percent of Subjects With Device Migration
Description: Longitudinal movement of all or part of the device for a distance ≥10 mm, as confirmed by CT scan, relative to anatomical landmarks and device positioning at the first post-operative CT scan
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 87
Participants | 0

22. Secondary Outcome: Percent of Subject With Thoracoabdominal Aneurysm (TAAA) Enlargement
Description: An increase in the maximum aneurysm diameter of 5 mm or more relative to the first post-operative CT scan within the 30 day follow-up window
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 93
Participants | 5

23. Secondary Outcome: Percent of Subjects With Severe Distal Thromboembolic Events
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 95
Participants | 2

24. Secondary Outcome: Percent of Subjects With Aortic Rupture
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 94
Participants | 1

25. Secondary Outcome: Percent of Subjects With Device or Procedure-related Laparotomy
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 95
Participants | 4

26. Secondary Outcome: Percent of Subjects With Conversion to Open Repair
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 94
Participants | 0

27. Secondary Outcome: Percent of Subjects With Aortoiliac Device Limb Occlusion
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 93
Participants | 0

28. Secondary Outcome: Percent of Subjects With Loss of Device Integrity
Description: Defined as any of the following:
  * Wire fracture identified in the sealing row stents of either the aortic, branch or iliac components
  * Transient (compression) or permanent stent-graft collapse (invagination) following complete device deployment, resulting in an overall reduction in the aortic, branch or iliac vessel luminal diameter
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 86
Participants | 14

29. Secondary Outcome: Percent of Subjects With Reintervention
Description: An additional unanticipated interventional or surgical procedure (including conversion to open surgery), related to the device (including withdrawal of the delivery system) or procedure.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 94
Participants | 15

30. Secondary Outcome: Percent of Subjects With Primary Patency
Description: Blood flow without occlusion maintained through the device after implant without an intervention. Assisted Primary Patency through 12 Months- Blood flow maintained through the device after implant regardless of re-interventions performed (without occlusion)
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 84
Participants | 61

31. Secondary Outcome: Percent of Subjects With Secondary Patency
Description: Blood flow through the device regardless of reinterventions performed (with or without occlusion) and freedom from surgical bypass
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 89
Participants | 79

32. Secondary Outcome: Percent of Subjects With Acute Kidney Injury
Description: >50% decrease in eGFR within 30 day follow-up window of TAMBE Device treatment when compared to pre-treatment serum creatinine value.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 91
Participants | 4

33. Secondary Outcome: Percent of Subjects With Renal Function Deterioration
Description: A sustained >25% decrease in eGFR over two consecutive study visits following TAMBE Device treatment when compared to pre-treatment serum creatinine value
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Study Arm
Number analyzed (Participants) | 74
Participants | 14

ADVERSE EVENTS:
Time Frame: 0-4 Years
Description: All subjects have not completed the 4 year follow-up, therefore the number and percentage of AEs may be under estimation of 4 year event rates.
Arm/Group | Primary Study Arm
All-Cause Mortality (participants affected / at risk) | 6/102
Serious Adverse Events (participants affected / at risk) | 52/102
Other Adverse Events (participants affected / at risk) | 92/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Study Arm (N=102)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Chronic anemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Symptomatic anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Acute decompensated heart failure (Cardiac disorders) | 1 (1)
Aortic valve insufficiency (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chronic atrial fibrillation (Cardiac disorders) | 1 (1)
Chronic systolic heart failure (Cardiac disorders) | 3 (3)
Congestive cardiac failure aggravated (Cardiac disorders) | 3 (5)
Congestive heart failure (Cardiac disorders) | 1 (1)
Congestive heart failure with acute exacerbation (Cardiac disorders) | 1 (1)
Ischemic cardiomyopathy (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 4 (4)
Non-sustained ventricular tachycardia (Cardiac disorders) | 1 (1)
Paroxysmal atrial fibrillation (Cardiac disorders) | 2 (2)
Systolic heart failure (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (2)
Bowel adhesions (Gastrointestinal disorders) | 1 (1)
Celiac artery stenosis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dysphagia aggravated (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2)
Hematochezia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal bleeding (Gastrointestinal disorders) | 3 (3)
Mesenteric arterial occlusion (Gastrointestinal disorders) | 1 (1)
Mesenteric artery stenosis (Gastrointestinal disorders) | 2 (2)
Mesenteric ischemia (Gastrointestinal disorders) | 1 (1)
Necrotizing pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis due to gallstones (Gastrointestinal disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Retroperitoneal hematoma (Gastrointestinal disorders) | 1 (1)
Short-bowel syndrome (Gastrointestinal disorders) | 1 (1)
Arterial stent occlusion (General disorders) | 2 (3)
Bare metal stent stenosis (General disorders) | 1 (1)
Calf swelling (General disorders) | 1 (1)
Endoleak (General disorders) | 1 (1)
Fever of unknown origin (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Renal stent-graft thrombosis (General disorders) | 1 (1)
Stent stenosis (General disorders) | 1 (1)
Stent thrombosis (General disorders) | 1 (2)
Stent-graft endoleak type IA (General disorders) | 1 (1)
Stent-graft endoleak type IC (General disorders) | 1 (1)
Stent-graft endoleak type II (General disorders) | 1 (1)
Unknown cause of death (General disorders) | 1 (1)
Vascular stent thrombosis (General disorders) | 1 (1)
Weakness generalized (General disorders) | 2 (2)
Acute cholecystitis (Hepatobiliary disorders) | 2 (2)
Bile duct stricture (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Liver cirrhosis (Hepatobiliary disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Aspiration pneumonia (Infections and infestations) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
COVID-19 respiratory infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Community acquired pneumonia (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2)
Hospital acquired pneumonia (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Prosthesis related infection (Infections and infestations) | 1 (1)
SARS-CoV-2 infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Femoral vein injury (Injury, poisoning and procedural complications) | 1 (1)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Volume overload (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower extremities weakness of (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenocarcinoma of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer of descending colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carcinoma in situ of breast ductal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant neoplasm of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Alzheimer's disease (Nervous system disorders) | 1 (1)
Brain lesion (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1)
Spinal cord ischemia (Nervous system disorders) | 4 (4)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1)
TIA (Nervous system disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (7)
Acute renal failure (Renal and urinary disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1)
End stage renal failure (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Kidney atrophy (Renal and urinary disorders) | 1 (1)
Renal artery dissection (Renal and urinary disorders) | 3 (3)
Renal artery occlusion (Renal and urinary disorders) | 2 (3)
Renal artery stenosis (Renal and urinary disorders) | 3 (3)
Renal artery thrombosis (Renal and urinary disorders) | 2 (2)
Renal infarction (Renal and urinary disorders) | 1 (1)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Acute on chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Aspiration pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Basilar atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Unilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical emphysema (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic rupture (Vascular disorders) | 1 (1)
Atheroembolism (Vascular disorders) | 1 (1)
Hemorrhagic shock (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
Popliteal artery thrombosis (Vascular disorders) | 1 (1)
Type A aortic dissection (Vascular disorders) | 1 (1)
Type B aortic dissection (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Study Arm (N=102)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Stent-graft endoleak type II (General disorders) | 59 (65)
COVID-19 (Infections and infestations) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Acute kidney injury (Renal and urinary disorders) | 7 (7)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator must wait until after the multi-center manuscript is published. Investigator will provide all Publications to allow the sponsor to review at least 60 days in advance of submission for publication or other public disclosure to suggest any modifications to protect proprietary information, and extend (as applicable) if filing a patent application.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT03728985/Prot_SAP_000.pdf